CLINICAL TRIAL: NCT03113344
Title: Population Pharmacokinetics of Anti-infective Drugs in Children in Anti-infectious Therapies
Brief Title: Population Pharmacokinetics of Anti-infective Drugs in Children With Infectious Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Shandong University (Other); Hopital Universitaire Robert-Debre (Other); Rennes University Hospital (Other)
Responsible Party: Principal Investigator, Adong Shen, Deputy Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Other Study IDs: BCH_PPK002; Yu-Jie Qi (Other: Beijing Children's Hospital); Wei Zhao (Other: Children's Hospital of Hebei Province；Shandong Provincial Qianfoshan Hospital); Hui Qi (Other: Beijing Children's Hospital); Fei Jin (Other: Beijing Children's Hospital); Evelyne Jacqz-Aigrain (Other: Robert Debre Hospital,Paris France); Stephanie Leroux (Other: Centre Hospitalier Universitaire de Rennes, France)
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Children; Infection
MeSH Terms: conditions — Infections | interventions — Cephalosporins; Antiviral Agents; Moxalactam; Ceftriaxone; Ceftazidime; Ampicillin; Penicillins; Amoxicillin; Erythromycin; Azithromycin; Meropenem; Imipenem; Ganciclovir; Acyclovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Biospecimen Retention: Samples With DNA — whole blood and plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with the usage of anti-infective drugs
  Interventions: Drug: cephalosporins,penicillins,macrolides,carbapenems and antiviral drugs

INTERVENTIONS:
Drug: cephalosporins,penicillins,macrolides,carbapenems and antiviral drugs — According to the models of population pharmacokinetics,the investigators and want to correlate use of antibiotics with treatment effectiveness and safety in children.
  Other Names: latamoxef; ceftriaxone; ceftazidime; ampicillin; penicillin; amoxicillin; erythromycin; azithromycin; meropenem; imipenem; ganciclovir; acyclovir

SUMMARY:
This study is based on the hypothesis that the pharmacokinetics of anti-infective drugs in children are different from adults. We aim to study the population pharmacokinetics of children receiving the anti-infective drugs for treatment of infectious diseases. In this study, we will detect drug concentration in plasma by using residual blood samples of blood gas analysis and other clinical tests and employ computers for constructing population pharmacokinetic models. In addition, we also want to correlate use of anti-infective drugs with treatment effectiveness and incidence of adverse effects in children. This novel knowledge will allow better and more rational approaches to the treatment of infectious diseases in children. It will also set the foundation for further studies to improve anti-infective drug therapies for children.

DETAILED DESCRIPTION:
1.Establish population pharmacokinetic (PPK) models of each anti-infective drug in children by nonlinear mixed effect modeling (NONMEM).

1. At different timepoint after antibiotic administration, plasma samples of 100 children will be collected from neonatal intensive care unit (NICU) and pneumology department for each drug. The clinical information includes demography, medication, concentration data, blood biochemical parameters and so on .
2. Plasma samples will be tested by high performance liquid chromatography (HPLC).
3. PPK models of antibiotics will be established by NONMEM program.
4. The reliability and stability of the PPK model will be evaluated by 1000 times of Bootstrap procedure and normalized predictive distribution error (NPDE).

2.Evaluation of the clinical feasibility and safety of individualized dosing.

1. According the results of PPK models, we will use dosages recommended in models to cure children infectious diseases in prospective studies. For each antibiotic, 50 children will be collected.
2. We will compare the therapeutic effects and safety between children with conventional therapies and children with individualized therapies, including proportions of children with effective drug concentration, improvement speed of of children, liver and kidney functions of of children, adverse reactions of drugs and so on.

ELIGIBILITY:
Inclusion Criteria:

* Children (0-18 years old) with anti-infective therapy against infectious diseases.
* The anti-infective therapy includes drugs commonly used in children infectious diseases, for example, cephalosporins (such as latamoxef, ceftazidime, ceftriaxone and so on), penicillins (such as penicillin, amoxicillin, ampicillin and so on), macrolides (such as erythromycin, azithromycin and so on), carbapenems (sucn as meropenem, imipenem and so on) and antiviral drugs (such as ganciclovir, acyclovir and so on).
* Children infectious diseases include pneumonia, sepsis, purulent meningitis and other diseases with infection.
* Informed consent signed by the parents and/or guardians.

Exclusion Criteria:

* Anti-infective drugs aren't involved in the therapies of children.
* It is unable to provide complete medical records or the current condition cannot accept the study process.
* Patients are allergic to anti-infective drugs.
* Parents and/or guardians do not agree to participate in this study.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with anti-infectious therapies.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-06-21 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum concentration (Cmax) | up to 4 weeks
  Cmax is a term used in pharmacokinetics refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose.

SECONDARY OUTCOMES:
time to achieve maximum concentration (Tmax) | up to 4 weeks
  Tmax is the term used in pharmacokinetics to describe the time at which the Cmax is observed.
absorption rate constant (ka) | up to 4 weeks
  Ka is the rate constant of drug absorption.
elimination rate constant (kel) | up to 4 weeks
  The elimination rate constant is a value used in pharmacokinetics to describe the rate at which a drug is removed from the system.
half-life (t1/2) | up to 4 weeks
  Half-life is the time required for a quantity to reduce to half its initial value.

CONTACTS AND LOCATIONS:
Overall Officials: A-Dong Shen, Master, Principal Investigator — Beijing Children's Hospital of Capital Medical University; Yu-Jie Qi, Master, Study Director — Beijing Children's Hospital of Capital Medical University; Wei Zhao, Doctor, Study Director — Children's Hospital of Hebei Province;Shandong Provincial Qianfoshan Hospital
Locations (1):
- Beijing Children's Hospital of Capital Medical University, Beijing, China

REFERENCES:
- [Result] Zhao W, Lopez E, Biran V, Durrmeyer X, Fakhoury M, Jacqz-Aigrain E. Vancomycin continuous infusion in neonates: dosing optimisation and therapeutic drug monitoring. Arch Dis Child. 2013 Jun;98(6):449-53. doi: 10.1136/archdischild-2012-302765. Epub 2012 Dec 19. PMID 23254142
- [Result] Leroux S, Zhao W, Betremieux P, Pladys P, Saliba E, Jacqz-Aigrain E; French Society of Neonatology. Therapeutic guidelines for prescribing antibiotics in neonates should be evidence-based: a French national survey. Arch Dis Child. 2015 Apr;100(4):394-8. doi: 10.1136/archdischild-2014-306873. Epub 2015 Jan 27. PMID 25628457
- [Result] Jacqz-Aigrain E, Leroux S, Zhao W, van den Anker JN, Sharland M. How to use vancomycin optimally in neonates: remaining questions. Expert Rev Clin Pharmacol. 2015;8(5):635-48. doi: 10.1586/17512433.2015.1060124. Epub 2015 Aug 4. PMID 26289222
- [Result] Ramos-Martin V, Johnson A, Livermore J, McEntee L, Goodwin J, Whalley S, Docobo-Perez F, Felton TW, Zhao W, Jacqz-Aigrain E, Sharland M, Turner MA, Hope WW. Pharmacodynamics of vancomycin for CoNS infection: experimental basis for optimal use of vancomycin in neonates. J Antimicrob Chemother. 2016 Apr;71(4):992-1002. doi: 10.1093/jac/dkv451. Epub 2016 Jan 10. PMID 26755499
- [Result] Zhao W, Hill H, Le Guellec C, Neal T, Mahoney S, Paulus S, Castellan C, Kassai B, van den Anker JN, Kearns GL, Turner MA, Jacqz-Aigrain E; TINN Consortium. Population pharmacokinetics of ciprofloxacin in neonates and young infants less than three months of age. Antimicrob Agents Chemother. 2014 Nov;58(11):6572-80. doi: 10.1128/AAC.03568-14. Epub 2014 Aug 25. PMID 25155587
- [Derived] Kan M, Shi HY, Han B, Wu YE, Li Q, Guo ZX, Li X, Hao GX, Zheng Y, Su LQ, Huang X, Sui ZG, Zhao W. Prediction of Unbound Ceftriaxone Concentration in Children: Simple Bioanalysis Method and Basic Mathematical Equation. Antimicrob Agents Chemother. 2020 Dec 16;65(1):e00779-20. doi: 10.1128/AAC.00779-20. Print 2020 Dec 16. PMID 33020163
- [Derived] Shi HY, Wang K, Wang RH, Wu YE, Tang BH, Li X, Du B, Kan M, Zheng Y, Xu BP, Shen AD, Su LQ, Jacqz-Aigrain E, Huang X, Zhao W. Developmental population pharmacokinetics-pharmacodynamics and dosing optimization of cefoperazone in children. J Antimicrob Chemother. 2020 Jul 1;75(7):1917-1924. doi: 10.1093/jac/dkaa071. PMID 32129861
- [Derived] Dong L, Zhai XY, Yang YL, Wang L, Zhou Y, Shi HY, Tang BH, Wu YE, Yang F, Wen L, Kong HX, Zhi LJ, Jacqz-Aigrain E, Zhao W. Population Pharmacokinetics and Dosing Optimization of Imipenem in Children with Hematological Malignancies. Antimicrob Agents Chemother. 2019 May 24;63(6):e00006-19. doi: 10.1128/AAC.00006-19. Print 2019 Jun. PMID 30962334
- [Derived] Dong Q, Leroux S, Shi HY, Xu HY, Kou C, Khan MW, Jacqz-Aigrain E, Zhao W. Pilot Study of Model-Based Dosage Individualization of Ganciclovir in Neonates and Young Infants with Congenital Cytomegalovirus Infection. Antimicrob Agents Chemother. 2018 Apr 26;62(5):e00075-18. doi: 10.1128/AAC.00075-18. Print 2018 May. PMID 29507070